CLINICAL TRIAL: NCT01349439
Title: Reduction of the Reconsolidation of the Trauma Memory With Propranolol
Brief Title: Reducing Reconsolidation of Trauma Memories With Propranolol
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Douglas Mental Health University Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Alain Brunet, Ph.D., Dr., Douglas Mental Health University Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 08-44
Record Dates: First submitted 2011-03-31; First posted 2011-05-06 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Propranolol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Propranolol + Memory Reactivation (Experimental): This arm involves recalling the traumatic event after administration of propranolol
  Interventions: Drug: Propranolol
- Placebo + Memory reactivation (Experimental): This arm involves recalling the traumatic event after administration of a placebo
  Interventions: Drug: Propranolol
- Placebo + No Memory Reactivation (Experimental): This arm involves administration of a placebo without recalling the traumatic event
  Interventions: Drug: Propranolol
- Propranolol + No Memory Reactivation (Experimental): This arm involves administration of propranolol without recalling the traumatic event
  Interventions: Drug: Propranolol
- Open-label Propranolol + Memory Reactivation (Other): All participants terminating the double-blind phase of the study will receive open-label reconsolidation blockade treatment with propranolol combined with recall of the traumatic event for six weeks.
  Interventions: Drug: Short acting + long acting propranolol + memory reactivation

INTERVENTIONS:
Drug: Propranolol — 1mg per Kg (participant weight)
  Arms: Placebo + Memory reactivation; Placebo + No Memory Reactivation; Propranolol + Memory Reactivation; Propranolol + No Memory Reactivation
Drug: Short acting + long acting propranolol + memory reactivation — After completing the double-blind phase of the study, participants will receive short acting propranolol 1mg/kg (patient weight) + long acting propranolol (1 or 1.5 mg/kg) followed by memory reactivation. Dose level for the long-acting propranolol will be randomly assigned across participants.
  Arms: Open-label Propranolol + Memory Reactivation

SUMMARY:
The purpose of this study is to test whether propranolol is capable of reducing subsequent physiological trauma-related conditioned responses, as well as self-reported post-traumatic stress disorder (PTSD) symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Suffer from chronic PTSD for at least 6 consecutive months;
* Obtain a score of 33 or more on the Impact of Events Scale-Revised:
* For participants aged 40 years: accept to undergo an electrocardiogram assessment. The results of the electrocardiogram must be normal;
* Accept to not commence taking new medications on a regular basis during the study.

Exclusion Criteria:

* Hypotension;
* Cardiac rhythm below 55 beats per minute;
* Medical conditions that contraindicates the administration of propranolol;
* Previous adverse reaction to, or non-compliance with, beta-blockers;
* Current use of medication that may involve potentially dangerous interactions with propranolol;
* Any medication that can have an impact on cardiac rhythm;
* Women who are breast feeding;
* Past or present bipolar disorder or psychosis,
* Present substance abuse or dependence, suicidal ideation;
* Participating in psychotherapy other than support psychotherapy;
* An average score above 20 on the Dissociative Experience Scale.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2011-03; Primary Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Electromyogram | Two weeks post-treatment
Heart rate | Two weeks post-treatment
Skin conductance | Two weeks post-treatment

SECONDARY OUTCOMES:
PTSD symptom levels | 2 to 26 weeks
  PTSD symptom levels will be assessed 2 to 26 weeks after randomization
Quality of life | 2 to 26 weeks
  Quality of life assessments will be conducted 2 to 26 weeks following randomization
Memory Experience | 2 to 26 weeks
  The Memory Experiences Questionnaire will be administered from 2 to 26 weeks following randomization
Psychophysiological assessments | 26 weeks
  Psychophysiological assessments will be repeated 26 weeks following randomization

CONTACTS AND LOCATIONS:
Overall Officials: Alain Brunet, Ph.D., Principal Investigator — Douglas Institute Research Centre
Locations (1):
- Douglas Mental Health University Institute, Verdun, Quebec, Canada

REFERENCES:
- [Background] Brunet A, Orr SP, Tremblay J, Robertson K, Nader K, Pitman RK. Effect of post-retrieval propranolol on psychophysiologic responding during subsequent script-driven traumatic imagery in post-traumatic stress disorder. J Psychiatr Res. 2008 May;42(6):503-6. doi: 10.1016/j.jpsychires.2007.05.006. Epub 2007 Jun 22. PMID 17588604